CLINICAL TRIAL: NCT02356809
Title: Safety and Efficacy Study of Pl-vegf165 to Treat Secondary Raynaud's Phenomenon Caused by Systemic Scleroderma
Brief Title: Safety and Efficacy Study of Gene Therapy Drug (Neovasculgen) to Treat Secondary Raynaud's Phenomenon
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Artgen Biotech (Other)
Collaborators: Russian Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAT
Record Dates: First submitted 2015-01-26; First posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-01

CONDITIONS: Secondary Raynaud's Phenomenon
Keywords: Gene therapy, plasmid, vegf, systemic scleroderma,secondary raynaud's phenomenon
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Systemic

ARMS (2):
- pl-vegf165 (Experimental): Patients of this group will receive 2,4 mg of pl-vegf165 administered by intramuscular injection which is given in the hand
  Interventions: Drug: Neovasculgen
- standard care (No Intervention): Patients of this group will receive standard therapy accepted in a clinical centre

INTERVENTIONS:
Drug: Neovasculgen — Neovasculgen is an original gene construction that contains supercoiled plasmid DNA (1.2 mg) that encodes pCMV-vegf165 as the active substance. The drug will be supplied to the study centre as a sterile lyophilisate that will be then dissolved in 2 ml of water for injections immediately prior to administration. The drug will be administered intramuscularly (interosseous muscles of hand) at 4-5 injection sites in the dorsal surface of the hand.
  Arms: pl-vegf165

SUMMARY:
The purpose of this study is to determine whether pl-vegf165 (Neovasculgen) is effective in the treatment of digital ulcers related to secondary Raynaud's phenomenon associated with systemic scleroderma

DETAILED DESCRIPTION:
This is a randomized, open, comparing clinical trial assessing the therapeutic efficacy of pl-vegf165 (Neovasculgen) in treating scleroderma-associated Raynaud's syndrome. Each patient of clinical group will undergo several intramuscular injections with a treatment dose of pl-vegf165 (Neovasculgen) in hand where digital ulcers locate. In the control group patients will receive only standard of care without gene therapy drug.

Study participants at the first study visit will complete study questionnaires, their hands will be assessed clinically for digital ulceration, and their hands will undergo non-invasive capillaroscopy. After this initial assessment, the patients of clinical group will undergo intramuscular injections of pl-vegf165 (Neovasculgen) in a hand altered with digital ulcers.

Patient will report the severity of their Raynaud's symptoms weekly over the six month study period. At three month post-injection, the patient will complete study questionnaires, their hands will be assessed clinically for digital ulceration, and their hands will undergo non-invasive capillaroscopy. At six months post-injection, the patient will again complete study questionnaires, their hands will be assessed clinically for digital ulceration, and their hands will undergo non-invasive capillaroscopy.

ELIGIBILITY:
Inclusion Criteria:

* obtained voluntary informed consent for participation in the clinical study
* presence of systemic scleroderma features satisfied to criteria of American College of Rheumatology classification
* presence at least one active digital ulcer at baseline

Exclusion Criteria:

* presence of another systemic connective tissue disease;
* absence at least one active digital ulcer at baseline;
* smoking within 3 months or smoking cessation using nicotine products;
* subjects currently taking sildenafil, tadalafil or vardenafil;
* history of sympathectomy over previous 12 months
* not able or unwilling to give voluntary informed consent for the study or follow requirements of the clinical study;
* decompensated chronic visceral diseases;
* clinically significant laboratory abnormalities;
* HIV, HBV and HCV antibodies in serum;
* alcohol or drug addiction;
* participation in other clinical studies (or administration of study products) within 3 months prior the study;
* conditions limiting study compliance (dementia, psycho-neurological diseases, drug addiction, alcoholism, etc.);
* malignancies including post-surgical period with chemo- and (or) radiation therapy);
* vascular malformations;
* pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of new digital ulcers | 180 days
  To determine the ability of pl-vegf165 to prevent development of new digital ulcers the frequency of new digital ulcers will be measured in both groups and then compared
Frequency of adverse events | 180 days

SECONDARY OUTCOMES:
Time of complete healing of digital ulcers | 180 days
  The ability of pl-vegf165 to accelerate the healing of the digital ulcer will be measured by estimating the area of the defect in progress
Pain scores on the visual analog scale | 180 days
  Visual analog scale is a diagnostic tool providing an assessment of the severity and quality of pain experienced by patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Stem Cell Institute, Moscow, Russia